CLINICAL TRIAL: NCT05049369
Title: Long-term Results of Tonsillectomy in the Treatment of Obstructive Sleep Apnea in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T205/2021
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Obstructive Sleep Apnea; Tonsillar Hypertrophy; Sleep Apnea Syndromes
Keywords: tonsillectomy; obstructive sleep apnea; tonsil surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polysomnography for all participants of the study (Experimental): Polysomnography device is used to measure certain variables overnight when a participant is sleeping
  Interventions: Device: Polysomnography

INTERVENTIONS:
Device: Polysomnography — Polysomnography is performed one time overnight

SUMMARY:
Long-term results of tonsillectomy in the treatment of obstructive sleep apnea in adults

DETAILED DESCRIPTION:
The investigators are studying long-term efficiency of tonsillectomy in adults with obstructive sleep apnea caused by tonsillar hypertrophy. These patients have undergone tonsillectomy in 2004-2018 and now 3-17 years later investigators will perform new polysomnographies and compare these results with preoperative values. Especially the reduction in apnea-hypopnea index (AHI) will be evaluated. The quality of life and possible symptoms will be measured with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* age at least 16 during tonsillectomy
* preoperative obstructive sleep apnea and AHI (apnea-hypopnea index) > 14
* tonsillectomy has been done because of the symptoms caused by tonsillar hypertrophy (ICD-10 diagnostic codes G47.3, R06.5 or J35.1)
* in addition to tonsillectomy, patients may have undergone shortening of uvula and/or radio frequency ablation of soft palate

Exclusion Criteria:

* AHI < 14
* in addition to tonsillectomy patient has undergone uvulectomy, uvulopalatoplasty, uvulopalatopharyngoplasty or mandibular advancement
* other, evaluated by investigator

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-04 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index | 3-17 years
  Post-operative apnea-hypopnea index (AHI) reduction by 50% compared to preoperative values in polysomnography.

SECONDARY OUTCOMES:
Quality of life measured by Glasgow Benefit Inventory (GBI) | 3-17 years
  General quality of life questionnaire. 18 questions, score 1-5 in each question, higher is better.
Quality of life measured by Epworth sleepiness scale (ESS) | 3-17 years
  Questions regarding sleepiness. Score 0-24, lower is better.
Apnea-index (AI) | 3-17 years
  Post-operative apnea index reduction compared to preoperative values in polysomnography.
Snoring time | 3-17 years
  Post-operative reduction of snoring time compared to preoperative values in polysomnography
Oxygen Desaturation Index (ODI) | 3-17 years
  Post-operative reduction of oxygen desaturation index compared to preoperative values in polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Jaakko M Piitulainen, MD,PhD, Principal Investigator — Department of Otorhinolaryngology, Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No